CLINICAL TRIAL: NCT00759785
Title: A Study to Establish Proof-of-Biology for MK-0646 in Breast Cancer
Brief Title: A Study of Dalotuzumab (MK-0646) in Breast Cancer Patients (MK-0646-013)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0646-013; MK-0646-013 (Other: Merck Registration Number); 2008-004180-18 (EudraCT Number)
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — dalotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ER-positive Luminal B (Experimental): Single dose of dalotuzumab 20 mg/kg infused intravenously over 60-120 minutes.
  Interventions: Drug: dalotuzumab (MK0646)
- Triple Negative (Experimental): Single dose of dalotuzumab 20 mg/kg infused intravenously over 60-120 minutes.
  Interventions: Drug: dalotuzumab (MK0646)

INTERVENTIONS:
Drug: dalotuzumab (MK0646) — Single intravenous infusion
  Other Names: MK-0646

SUMMARY:
A study to evaluate the response of growth factor signatures (GFS) to a single dose of dalotuzumab in participants with triple negative (TN) or estrogen receptor (ER)-positive luminal B breast cancer. The primary hypothesis is that dalotuzumab will induce a decrease in the GFS in at least 40% of participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant has operable stage I-IIIa breast cancer of the following subtypes: (1) estrogen receptor (ER)-negative, progesterone receptor (PR)-negative, and human epidermal growth factor receptor 2 (HER2)-negative breast cancer; (2) ER-positive tumor meeting one of the following criteria: histologic grade 3; histologic grade 2 and PR-negative; histologic grade 2 and Ki67 antigen ≥10%. Tumor is at least 2 cm in diameter as assessed by physical or radiographic exam
* Participant is female and ≥18 years of age

Exclusion Criteria:

* Participant is pregnant, breastfeeding or planning to become pregnant while in the study
* Participant has received prior chemotherapy, biological therapy or radiation
* Participant has participated in a clinical trial in the last 30 days
* Participant has a history of drug or alcohol abuse in the last year
* Participant is human immunodeficiency virus (HIV) positive. Patient has a history of Hepatitis B or C
* Participant has poorly controlled diabetes mellitus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-09-30 (Actual); Primary Completion 2010-02-17 (Actual); Study Completion 2010-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- ER-positive Luminal B (ER+): ER-positive Luminal B participants received a single dose of dalotuzumab 20 mg/kg infused over 60-120 minutes.
- Triple Negative (TN): Triple Negative participants received a single dose of dalotuzumab 20 mg/kg infused over 60-120 minutes.
Period: Overall Study
Arm/Group | ER-positive Luminal B (ER+) | Triple Negative (TN)
Started | 26 | 22
Treated | 25 | 20
Completed | 14 | 17
Not Completed | 12 | 5
Not completed — Participant sample not evaluable | 11 | 2
Not completed — Participant sample lost | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ER-positive Luminal B (ER+) | Triple Negative (TN) | Total
Number analyzed (Participants) | 26 | 22 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.8 (15.7) [30 to 91] | 55.1 (14.1) [32 to 57] | 57.1 (14.9) [30 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Demonstrating a Decrease in the Growth Factor Signature (GFS)
Description: GFS was measured by microarray analysis of the entire 101 gene signature expression. The GFS is quantified as the change in gene expression between two separate samples collected from the same participant. A log (base 10) ratio of expression in the post-dose sample was generated relative to the reference in both the Up and DOWN arms of the gene signature. A log ratio value of zero indicated no change in the expression between the two samples. GFS was calculated as the mean log ratio of genes in the UP arm minus mean log ratio of genes in the Down arm. GFS was compared for paired samples (pre-dose and post-dose) by a T-statistic calculated as the GFS divided by its standard error. Responders to therapy had a T-statistic that was smaller than the threshold 1st percentile of student's T-distribution and were counted as having a decrease in GFS.
Time Frame: Up to 12 Days Post-dose
Population: All participants who received a single dose of dalotuzumab and had evaluable baseline and post-dose biopsy samples.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | ER-positive Luminal B (ER+) | Triple Negative (TN)
Number analyzed (Participants) | 14 | 17
Percentage of participants | 28.6 [13.1 to 49.2] | 17.6 [6.7 to 35.2]

2. Secondary Outcome: Percentage of IGF1R Positive Participants With a Decrease in GFS by Cohort
Description: Insulin-like Growth Factor Receptor Type 1 (IGF1R) expression was measured in pre-dose biopsy samples using an immunohistochemistry assay to establish baseline IGF1R positivity. Biopsy samples were considered IGF1R positive if at least 10% of tumor cells stain with intensity 1+ or greater based on staining criteria of very weak (+/-); weak (1+); moderate (2+); or strong (3+). GFS response was correlated with IGF1R expression for ER-positive luminal B and triple negative cohorts.
Time Frame: Up to 12 Days Post-dose
Population: All participants who received a single dose of dalotuzumab, were IGF1R positive at baseline, and had evaluable postdose biopsy samples.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | ER-positive Luminal B (ER+) | Triple Negative (TN)
Number analyzed (Participants) | 12 | 9
Percentage of participants | 25.0 [9.6 to 47.5] | 11.1 [1.2 to 36.8]

3. Secondary Outcome: Percentage of IGF1R Negative Participants With a Decrease in GFS by Cohort
Description: Biopsy samples were considered IGF1R negative if less than 10% of tumor cells stain. GFS response was correlated with IGF1R expression for ER-positive luminal B and triple negative cohorts.
Time Frame: Up to 12 Days Post-dose
Population: All participants who received a single dose of dalotuzumab, were IGF1R negative at baseline, and had evaluable postdose biopsy samples.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | ER-positive Luminal B (ER+) | Triple Negative (TN)
Number analyzed (Participants) | 1 | 5
Percentage of participants | 0.0 [0.0 to 90.0] | 20.0 [2.1 to 58.4]

4. Secondary Outcome: Change From Baseline in IGF1R Membrane H-Score After a Single Dose of Dalotuzumab
Description: IGF1R expression was measured in pre and post-dose biopsy samples using an immunohistochemistry assay. Results were expressed as an IGF1R membrane H-score. The H-score was calculated from the percentage of cells staining very weak (+/-); weak (1+); moderate (2+); or strong (3+) and obtained by the formula: (3 x percentage of strongly staining nuclei) + (2 x percentage of moderately staining nuclei) + (1 x percentage of weakly staining nuclei) + (0.5 x percentage of weakly staining nuclei). The H-score ranges from 0 to 300; with a score of 0 representing the absence of IGF1R expression and an H-score of 300 representing maximum IGF1R expression. A decrease in IGF1R membrane H-score was an indication of target engagement by dalotuzumab. A larger decrease in H-score correlated with a greater target engagement
Time Frame: Baseline and Up to 12 Days
Population: All participants who received a single dose of dalotuzumab, had evaluable baseline and post-dose biopsy samples, and had H-score data available for pre- and post-dose measurements.
Measure: Mean (Full Range); unit: H-score
Arm/Group | ER-positive Luminal B (ER+) | Triple Negative (TN)
Number analyzed (Participants) | 13 | 13
H-score | -104.5 [-235 to -4] | -11.5 [-105 to 100]

ADVERSE EVENTS:
Time Frame: Up to 12 Days Post-dose
Description: Adverse events for all participants who received a single dose of dalotuzumab
Arm/Group | ER-positive Luminal B (ER+) | Triple Negative (TN)
Serious Adverse Events (participants affected / at risk) | 1/25 | 1/20
Other Adverse Events (participants affected / at risk) | 2/25 | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ER-positive Luminal B (ER+) (N=25) | Triple Negative (TN) (N=20)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1)
Breast cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ER-positive Luminal B (ER+) (N=25) | Triple Negative (TN) (N=20)
Nausea (Gastrointestinal disorders) | 1 (2) | 4 (5)
Fatigue (General disorders) | 1 (1) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation and can delete information identified as confidential prior to submission.